CLINICAL TRIAL: NCT02950792
Title: A Study of Adaptive Radiotherapy Using ViewRay MRI Based Imaging in Locally Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: MRI Adaptive Replanning Using ViewRay
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator Decision
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Adrian Ishkanian, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160397
Record Dates: First submitted 2016-10-24; First posted 2016-11-01 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; Spermine Synthase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ViewRay MRI-IGART (Experimental): ViewRay MRI-Image-Guided Adaptive Radiation Therapy (IGART):
  * Daily MRI on ViewRay 5 days per week for 4 weeks in combination with weekly standard of care chemo-radiation.
  * Daily MRI on ViewRay during Week 5 in combination with Stereotactic Body Radiation Therapy boost for daily for up to 1 week.
  * Continued standard of care consolidation chemotherapy every 21 days for 3 cycles, beginning 4 - 6 weeks after completion radiation therapy, .
  Interventions: Device: ViewRay MRI; Radiation: Stereotactic Body Radiation Therapy Boost

INTERVENTIONS:
Device: ViewRay MRI — ViewRay Magnetic Resonance Imaging
  Other Names: ViewRay Magnetic Resonance Imaging
Radiation: Stereotactic Body Radiation Therapy Boost — In the (week 5), all patients will have a week 5 MRI and Four-dimensional computed tomography (4D CT) for purposes of planning Phase II boost. Gross tumors < 5 cm will receive a MR-based adaptive replanning Stereo boost of 80 Gy - 90 Gy (20 Gy-30 Gy in 5 fractions). Gross tumors < 5cm will receive an MR-based adaptive replan fractionated boost to 74 Gy at 2.4 Gy/day. Individualized radiation therapy prescription to primary tumor will maintain organs at risk (OAR) constraints to lung including mean lung dose (MLD) < 20 Gy with V20 < 37%. Simultaneously, MRI-based adaptive replanning boost of 12 Gy in 5 fractions (2.4 Gy/day) will be given to gross lymph nodes. Final doses prescribed will be limited by doses to all OARs.
  Other Names: Stereotactic radiosurgery (SRS) Boost

SUMMARY:
Current dose escalation regimens with and without chemotherapy have failed to achieve improved local control and overall survival over standard of care therapy to date. Difficulties with dose escalation have been largely due to dose limiting toxicities of surrounding normal organs, in particular to the normal lung parenchyma, and esophagus. Real time, online adaptive planning using magnetic resonance imaging (MRI) could achieve significant volume reduction of primary lung disease over the course of therapy, thereby reducing dose to normal structures, and providing a mechanism in which to dose escalate safely, and more effectively with accurate target delineation.

The investigators hypothesize that MRI based adaptive planning will provide a novel method to dose escalate safely with acceptable organ at risk doses. In addition, further improvements in radiotherapy targeting accuracy, normal tissue avoidance, and conformality of target-tissue coverage will be achieved through the use of 4D real-time tracking which is derived by deformably registering daily MR and planning MR (MRsim) and Computed Tomography Simulator (CTsim) with advanced non-rigid image-registration tools.

DETAILED DESCRIPTION:
This study is a single-arm phase II study of adaptive radiotherapy using ViewRay MRI based imaging in locally Advanced non-small cell lung cancer patients. Randomization is not applicable.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have primary lung tumor identified on MRI, histologically proven to be NSCLC.
2. Patients must be clinical AJCC stage IIIA or IIIB (AJCC 7th ed) with non-operable disease; evaluated by a multidisciplinary treatment team including at least 1 thoracic surgeon within 8 weeks prior to registration.
3. Patients with multiple, ipsilateral pulmonary nodules (T3, or T4) are eligible
4. Minimum diagnostic workup to include:

   * History/physical examination, including documentation of weight, within 8 weeks prior to registration (2 weeks optimal)
   * Diagnostic CT scan for staging and RT plan within 4 weeks prior to registration;
   * CT scan or sim CT of chest and upper abdomen (IV contrast is recommended unless medically contraindicated) within 6 weeks prior to registration;
   * CT scan of the brain (contrast is recommended unless medically contraindicated) or MRI of the brain within 6 weeks prior to registration
   * Able to tolerate repeated MRI imaging
   * Pulmonary function tests, including diffusing capacity of the lung for carbon monoxide (DLCO), within 6 weeks prior to registration; patients must have forced expiratory volume in one second (FEV1) ≥ 1.2 Liter or ≥ 50% predicted without bronchodilator;
   * Zubrod Performance Status 0-1 within 2 weeks prior to registration
   * Age ≥ 18;
   * Complete blood count (CBC)/differential obtained no more than 8 weeks prior to registration on study, with adequate bone marrow function defined as follows:

     * White blood cell (WBC) ≥ 4000/ml
     * Absolute neutrophil count (ANC) ≥1,800 cells/mm
     * Platelets ≥100,000 cells/mm
     * Hemoglobin ≥ 10.0 mg/dl (Note: the use of transfusion or other intervention to achieve this level is acceptable)
   * Serum creatinine, blood urea nitrogen, alanine aminotransferase (ALT), aspartate aminotransferase (AST), Alk Phos, total bilirubin, serum electrolytes (eg. Sodium, potassium, chloride, bicarbonate, calcium), glucose, total protein, albumin will be drawn no greater than 8 weeks prior to enrollment.

     * Serum creatinine of 1.5mg or less; serum bilirubin of 2.0mg or less; creatinine clearance of 60ml/min or greater no more than 4 weeks prior to registration (Note: calculated creatinine clearance is permissible. If the creatinine clearance is greater than 60ml/min, then a serum creatinine of up to 1.8mg is allowable at the discretion of the PI
   * Serum pregnancy test for female patients of childbearing potential, ≤8 weeks prior to enrollment; women of childbearing potential and male participants must practice adequate contraception on trial
   * Patients must be able to provide study-specific informed consent prior to study entry
   * Patients must agree to have their biopsy tissue and blood banked for future molecular studies

Exclusion Criteria:

1. Patients with any component of small cell lung carcinoma are excluded
2. Evidence of distant metastases.
3. Patients with evidence of a malignant pleural or pericardial effusion.
4. Previous systemic chemotherapy (for any cancer) or pelvic radiation therapy
5. A prior or concurrent malignancy of any other site or histology unless the patient has been disease free for greater than or equal to five years except for nonmelanoma skin cancer and/or stage T1a prostate cancer or carcinoma in situ of the uterine cervix.
6. Prior radiotherapy that would result in overlap of radiation fields
7. Patients taking drugs with potential nephrotoxicity or ototoxicity (such as aminoglycosides)
8. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
9. Prior allergic reaction to the study drug(s) involved in this protocol
10. Patients with T4 disease with radiographic evidence of invasion of a large pulmonary artery and tumor causing significant narrowing and destruction of that artery are excluded.
11. Severe active co-morbidity:

    * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
    * Transmural myocardial infarction within the last 6 months
    * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
    * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
    * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects (Note: laboratory tests for liver function and coagulation parameters are not required for entry into this protocol)
    * Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition (Note: HIV testing is not required for entry into this protocol) The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immune-compromised patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08 (Estimated); Primary Completion 2017-08-08 (Actual); Study Completion 2017-08-08 (Actual)

PRIMARY OUTCOMES:
Rate of Locoregional Failure/Progression (LRF/LRP) in Study Participants Receiving Protocol Therapy. | Up to 2 Years After Protocol Therapy
  MRI-based adaptative radiation planning can provide a method for dose escalation to improve locoregional Failure (LRF/LRP) rates at 2 years in study participants. Locoregional failure/progression (LRF/LRP) will be defined as development of progressive lung cancer centered within 1 cm from the initial planning target volume (PTV). Progressive disease in any of the 14 nodal stations will be considered as regional recurrence. Progression will be assessed by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria. with integration of MRI/CT.
Rate of Severe Treatment-Induced Toxicity | Up to 2 Years Post-End of Protocol Therapy
  Rate of severe (grade 3 CTCAE, v.4) radiation-induced lung toxicity (RILT) and other severe adverse events, including grade 3+ (CTCAE, v.4) esophagitis, or grade 2 pericardial effusions, or any grade cardiac adverse events related to chemo-radiation using MRI-based adaptive planning vs. historical controls using conventional plans.

SECONDARY OUTCOMES:
Rate of Overall Survival (OS) in Study Participants | Up to 3 years after protocol therapy.
  Rate of overall survival in study participants using MRI-based adaptive planning vs historical controls. Overall survival is defined as the length of time from the start of treatment that study participants are still alive.
Rate of Progression-Free Survival (PFS) in Study Participants | Up to 3 years after protocol therapy.
  Rate of progression-free survival in study participants using MRI-based adaptive planning vs historical controls. Progression-Free Survival (PFS) is defined as the length of time that passes from the start date of protocol therapy until the date on which disease "progresses" or the date on which the participant dies, from any cause. Disease progression will be assessed using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria.
Rate of Lung Cancer-Specific Survival | Up to 3 years after protocol therapy.
  Rate of Lung Cancer-specific survival in study participants using MRI-based adaptive planning vs historical controls. Lung cancer-specific survival is defined as the length of time that passes from the date of diagnosis or start date of protocol therapy until the date of death from lung cancer.
Comparison of Gross Tumor Volumes (GTV) defined by MRI vs. FanBeam CT (FBCT) at CT Simulation and at each adaptive planning time point. | Daily Up to 5 weeks after start of protocol therapy
  Gross tumor volumes (GTVs) at a specific time point between MRI and Fan Bean CT will be compared using Mann-Whitney test.
Development of a Database consisting all Daily MR data sets to support further research. | Up to 5 years
  Potential applications include determination of optimal adaptive planning frequency and the benefits of basing IGART on 4D anatomic datasets derived from deformably registering daily MR and planning FBCT and MR datasets.
Predictivity of Volumetric Changes in MRI Imaging for Locoregional failure/progression (LRP) and Organs at Risk (OARs) toxicity. | Up to 5 years
  Predictivity of volumetric changes in MRI imaging for LRP and OAR toxicity will be assessed using time-dependent receiver operating characteristic (ROC) method and regular ROC method, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Ishkanian, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States